CLINICAL TRIAL: NCT04205851
Title: An Ascending Single- and Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneous Gimsilumab in Healthy Subjects and Subjects With Ankylosing Spondylitis
Brief Title: Phase 1 Study With KIN-1901 in Healthy Subjects and Subjects With Ankylosing Spondylitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kinevant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KIN-1901-1001
Record Dates: First submitted 2019-12-04; First posted 2019-12-20 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Inflammation; Rheumatic Diseases
Keywords: Spondylitis, Ankylosing
MeSH Terms: conditions — Inflammation; Rheumatic Diseases; Spondylitis, Ankylosing | interventions — gimsilumab

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind (Sponsor unblind), multi-cohort, placebo-controlled design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- KIN-1901 (Experimental): Single or repeat (once weekly for 4 weeks) KIN-1901 subcutaneous injection
  Interventions: Drug: KIN-1901
- Placebo (Placebo Comparator): Single or repeat (once weekly for 4 weeks) placebo subcutaneous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KIN-1901 — KIN-1901 is a fully human monoclonal antibody (mAb).
  Arms: KIN-1901
Drug: Placebo — Saline
  Arms: Placebo

SUMMARY:
This study is intended to treat ankylosing spondylitis (AS). AS is a form of arthritis that primarily affects the spine. It is characterized by inflammation of the spinal joints that can lead to severe pain, and in more advanced cases, ankylosis (sections of the spine fuse in a fixed, immobile position). The study will be an ascending single and multiple-dose study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of subcutaneous KIN-1901 in healthy subjects and subjects with AS.

DETAILED DESCRIPTION:
KIN-1901 is a fully human immunoglobulin monoclonal antibody (mAb) directed towards a proinflammatory cytokine that is believed to have a role in inflammation and autoimmunity, and is found in synovial fluid from patients with spondyloarthritis. Therefore, neutralization of this cytokine activity by specific monoclonal antibodies (mAbs) could be beneficial in treating certain spondyloarthropathies such as ankylosing spondylitis (AS).

The primary objective of the study is to evaluate the safety and tolerability of escalating single-dose or once-weekly repeat-dose subcutaneous (SC) administration of KIN-1901 in healthy subjects (Cohorts 1 through 4) and in subjects with AS (Cohort 5). The secondary objective of the study is to evaluate the pharmacokinetics (PK) of escalating single-dose and once-weekly repeat-dose SC administration of KIN-1901 in healthy subjects (Cohorts 1 through 4) and in subjects with AS (Cohort 5). The following exploratory objectives will also be evaluated: (1) To explore the pharmacodynamic (PD) effects of escalating single-dose and once-weekly repeat-dose SC administration of KIN-1901 in healthy subjects (Cohorts 1 through 4), (2) To explore the PD effects and changes in disease activity by Assessment in Ankylosing Spondylitis Criteria ASAS 20/40 (and components) and Ankylosing Spondylitis Disease Activity Score-CRP (ASDAS-CRP) of once-weekly repeat-dose SC administration of KIN-1901 in subjects with AS (Cohort 5), (3) To assess biomarkers of efficacy and safety after once-weekly repeat-dose SC administration of KIN-1901 in subjects with AS (Cohort 5).

ELIGIBILITY:
Main Inclusion Criteria:

1. Capable of giving written informed consent, which includes compliance with study requirements and restrictions listed in the consent form.
2. Age requirements:

   * Cohorts 1 through 4 (healthy): Male or female age ≥ 18 years and ≤ 50 years.
   * Cohort 5 (AS): Male or female age ≥ 18 years and ≤ 75 years.
3. Females must agree to use a highly effective birth control method (<1% failure rate per year) throughout the study, reproductive status of non-childbearing based on medical history, or is postmenopausal:

   * Non-childbearing potential defined as pre-menopausal female with medical history of bilateral tubal ligation, bilateral oophorectomy (removal of the ovaries) or hysterectomy; hysteroscopic sterilization,
   * Postmenopausal defined as 12 months of spontaneous amenorrhea; with follicle stimulating hormone (FSH) confirmation.
   * Woman of Childbearing potential (WCBP) who is already using an established method of highly effective contraception or agrees to use one of the allowed BC methods for at least 28 days prior to the start of dosing (as determined by the Investigator Brochure or Investigator or designee) to sufficiently minimize the risk of pregnancy throughout study participation (until completion their study follow-up visit).
4. Males who are sexually active must agree to use one of the allowed birth control methods. Male subjects must also agree to sufficiently minimize the risk of pregnancy throughout study participation (until completion their follow-up visit).
5. Body Mass Index (BMI):

   * Cohorts 1-4 (healthy): BMI 18.5 to 31 kg/m2 at Screening
   * Cohort 5 (AS): BMI 18 to 33 kg/m2 at Screening

   Additional Inclusion Criteria for Cohort 5 (AS) only:
6. AS diagnosis fulfilling the Modified New York criteria for AS.
7. Active AS, as defined by the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) ≥ 4 despite NSAID, corticosteroid or DMARD therapy.
8. BASDAI, item 2, spinal pain score ≥ 4 (out of 10).
9. AS diagnosis confirmed by Sacroiliac (SI) imaging within the last 2 years (confirmed by central reader during Screening).
10. Does not have a history of complete spinal ankylosis.
11. CRP > ULN at Screening.
12. Two prior failures to NSAID therapy (sub-optimal clinical response following four weeks at maximum tolerated dose) or intolerance to NSAID therapy.

Main Exclusion Criteria:

An individual will NOT be eligible for inclusion in this study if any of the following criteria apply.

1. Clinically significant illness which required medical treatment within 8 weeks or a clinically significant infection within 4 weeks prior to Screening.
2. Disease diagnosis that may influence the outcome of the study; such as psychiatric disorders or disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, cardiovascular system within 4 weeks prior to randomization, or individuals who have preexisting metabolic congenital abnormality(ies).
3. Positive Quantiferon test.
4. Use of prescription and non-prescription drugs:

   * Cohorts 1 through 4 (healthy): Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 14 days or 5 half-lives (whichever is longer) prior to the first dose of study treatment, unless in the opinion of an Investigator and Medical Monitor the medication will not interfere with the study procedures or compromise subject safety or permitted under Section 5.10.1.
   * Cohort 5 (AS):
   * Current or prior treatment regimen that includes a biologic therapy (e.g., anti-TNF-alpha, anti-IL-17A, anti-IL-6, or anti-IL-12/23)
   * Use of parenteral and/or intra-articular steroids or immunosuppressants within 6 weeks prior to the first dose of study treatment.

   Oral steroids are permitted if the dosage is ≤10 mg/day prednisone (or equivalent) and is stable for a minimum of 4 weeks before the first dose of study treatment and remains unchanged throughout the study.

   Also note:

   Oral NSAID treatment is permitted if the dosage is stable for a minimum of 2 weeks before the first dose of study treatment and remains unchanged throughout the study.

   Oral sulfasalazine treatment is permitted if the dosage is ≤ 3 g/d (max) and is stable for a minimum of 4 weeks before the first dose of study treatment and remains unchanged throughout the study.

   Oral methotrexate use is permitted if used for a minimum of 3 months, the dosage is ≤ 20 mg/week, and is the dose stable for a minimum of 4 weeks (including dosage of concomitant folate) before the first dose of study treatment and remains unchanged throughout the study.

   Subcutaneous methotrexate use is permitted if the dosage is ≤ 20 mg/week and is stable for a minimum of 4 weeks (including dosage of concomitant folate) before the first dose of study treatment and remains unchanged throughout the study.
5. Individual who received an investigational product (including placebo) 30 days prior to the start of dosing (5 half-lives or twice the duration of the biological effect of the investigational product), whichever is longer.
6. Weight loss or gain of >10% between screening and up to the start of dosing.
7. Hemoglobin level ≤ 12 g/dL at Screening.
8. Positive result for HIV (HIV-1/HIV-2 Antibodies), HBsAg or HCVAb screening tests.
9. Known or suspected history of drug abuse (amphetamines, barbiturates, cannabinoids, cocaine, opiates and phencyclidine) or alcohol misuse* within 6 months prior to Screening, or a positive urine drug test and/or alcohol breathalyzer test at Screening or baseline.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2020-04-07 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | Up to 57 days (Cohort 1 and 2); Up to 78 days (Cohorts 3, 4, and 5)
Change from baseline in QTcF interval | Up to 57 days (Cohort 1 and 2); Up to 78 days (Cohorts 3, 4, and 5)
Change in clinical chemistry parameter hsCRP determined by laboratory testing | Up to 57 days (Cohort 1 and 2); Up to 78 days (Cohorts 3, 4, and 5)
Incidence of serum anti-drug antibodies | Up to 57 days (Cohort 1 and 2); Up to 78 days (Cohorts 3, 4, and 5)

SECONDARY OUTCOMES:
Serum Cmax | Up to 57 days (Cohort 1 and 2); Up to 78 days (Cohorts 3, 4, and 5)
  Maximum observed concentration
Serum tmax | Up to 57 days (Cohort 1 and 2); Up to 78 days (Cohorts 3, 4, and 5)
  Time to Cmax
Serum AUC | Up to 57 days (Cohort 1 and 2); Up to 78 days (Cohorts 3, 4, and 5)
  Area under the concentration-time curve

CONTACTS AND LOCATIONS:
Locations (1):
- Altasciences Clinical Research, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No